CLINICAL TRIAL: NCT04387513
Title: Impact of Cardiac Surgery in Severe Left Endocarditis With Neurological Complications: a Multicentric,Retrospective, Propensity-score Matching Study
Brief Title: Impact of Early Cardiac Surgery in Severe Left Endocarditis With Neurological Complications: a Retrospective Study
Acronym: ICE-COCA
Status: Completed | Type: Observational
Sponsor: Gros, Alexandre, M.D. (Individual)
Responsible Party: Principal Investigator, Dr Alexandre Gros, GROS, Alexandre, Medical Doctor, Intensive Care Unit, Principal Investigator, Gros, Alexandre, M.D.
Other Study IDs: AlexandreGros
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Endocarditis; Neurologic Complication
MeSH Terms: conditions — Endocarditis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac surgery — Cardiac surgery, if indicated, delayed or not by neurological complications

SUMMARY:
Surgical delay in severe endocardits, with neurological complications, is still debated. Early surgery, if indicated, permits to avoid new embolic events, or to fix valvular damages, but can create or increase a cerebral hemorrage.

Hypothesis Cardiac surgery, as soon as possible, if indicated, would reduce mortality, in severe left endocarditis, with neurological complications.

Primary objective To assess the impact of early versus late cardiac surgery on mortality at 1 year, in patients with severe endocarditis, with neurological complications.

Primary endpoint:

1) Mortality at 1 year

Secondary endpoints:

1. Analyze the factors associated with neurological degradation
2. Evaluate the neurological tolerance of cardiac surgery.

DETAILED DESCRIPTION:
Surgical delay in severe endocardits, with neurological complications, is still debated. Early surgery, if indicated, permits to avoid new embolic events, or to fix valvular damages, but can create or increase a cerebral hemorrage.

Hypothesis Cardiac surgery, as soon as possible, if indicated, would reduce mortality, in severe left endocarditis, with neurological complications.

Primary objective To assess the impact of early versus late cardiac surgery on mortality at 1 year, in patients with severe endocarditis, with neurological complications.

Primary endpoint:

1) Mortality at 1 year

Secondary endpoints:

1. Analyze the factors associated with neurological degradation
2. Evaluate the neurological tolerance of cardiac surgery.

Methods Multicentric study (7 French university hospitals). Retrospective study: from august 2010 to december 2017. Propensity score matching study. 192 patients are included.

ELIGIBILITY:
Inclusion Criteria:

* Left endocarditis
* With indication of cardiac surgery
* Severe endocaditis (SOFA score > or = 3/16)
* With pre operative neurological complications

Exclusion Criteria:

* Age < 18
* Right endocarditis without left endocarditis
* No severe endocarditis (SOFA score < 3)
* Ne pre operative neurological complications
* Endocarditis without indication of cardiac surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in intensive care unit. They all have an indication of surgery, but they are not all operated (neurological or others contre-indications).
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2010-08-18 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | at 1 year after the diagnosis of endocarditis
  Death from any cause

SECONDARY OUTCOMES:
Neurogical tolerance | At 6 months
  Modified Rankin score after cardiac surgery, 0 (no symptoms at all) to 6 (death)

IPD SHARING:
Plan to Share IPD: Undecided
All individual data are available in an Excel file.